CLINICAL TRIAL: NCT01338610
Title: Evaluation of ESBA105 in the Persistent Relief of Ocular Discomfort in Patients With Severe Dry Eye
Brief Title: ESBA105 in Patients With Severe Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-079
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Eyes Dry Chronic
Keywords: Ocular discomfort
MeSH Terms: interventions — ESBA105

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESBA105 (Experimental): ESBA105 ophthalmic solution, 1 drop in each eye 3 times per day for 4 weeks
  Interventions: Biological: ESBA105 ophthalmic solution
- Vehicle (Placebo Comparator): ESBA105 vehicle, 1 drop in each eye 3 times per day for 4 weeks
  Interventions: Other: ESBA105 vehicle

INTERVENTIONS:
Biological: ESBA105 ophthalmic solution
  Arms: ESBA105
Other: ESBA105 vehicle — Inactive ingredients used as Run-In and placebo comparator
  Arms: Vehicle

SUMMARY:
The purpose of this study was to evaluate the efficacy of ESBA105 over vehicle in reducing the ocular symptoms of dry eye disease, as measured by a mean global Visual Analog Scale (VAS) discomfort score.

DETAILED DESCRIPTION:
Following Run-In, patients qualifying for treatment were randomized 2:1 to receive ESBA105 (experimental group) or Vehicle (control group) for 4 weeks. Patients not qualifying for treatment (based on global VAS discomfort score), were discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing physician diagnosis of dry eye for at least 6 months.
* Use of artificial tears, gels, lubricants, or re-wetting drops on a regular basis.
* Experience persistent ocular discomfort.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Contact lens wearers.
* Severe Sjogren's Syndrome.
* History of corneal surgery including refractive surgeries.
* Intraocular surgery within 6 months of Visit 1.
* Intraocular or periocular injection within 6 months of Visit 1.
* Lid function abnormalities.
* Use of steroids, tetracycline, doxycycline, etc., within 30 days of Visit 1.
* Any acute infectious or non-infectious ocular condition of the anterior or posterior segments in either eye within 30 days of Visit 1.
* Diseases/conditions of ocular surface associated with clinically significant scarring/destruction of conjunctiva/cornea.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 16 investigative sites located within the United States. Participant flow data is presented for all subjects exposed to product.
Pre-assignment Details: Of the 334 enrolled, 210 subjects did not qualify for Run-In and were exited from the study without exposure to product. Of the 124 entering Run-In, 39 did not qualify for treatment. The 85 subjects qualifying for treatment were randomized 2:1 to receive either ESBA105 or Vehicle.
Groups:
- Run-In Only: ESBA105 vehicle
- ESBA105: ESBA105 vehicle (Run-In), ESBA105 ophthalmic solution (treatment)
- Vehicle: ESBA105 vehicle (Run-In), ESBA105 vehicle (treatment)
Period: Overall Study
Arm/Group | Run-In Only | ESBA105 | Vehicle
Started | 39 | 56 | 29
Completed | 34 | 55 | 28
Not Completed | 5 | 1 | 1
Not completed — Patient Decision Unrelated to Advs Event | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Adverse Event | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data is presented for all subjects exposed to product.
Groups:
- ESBA105: ESBA 105 vehicle (Run-In), ESBA105 ophthalmic solution (treatment)
- Total: Total of all reporting groups
Arm/Group | Run-In Only | ESBA105 | Vehicle | Total
Number analyzed (Participants) | 39 | 56 | 29 | 124
Age, Customized [Number; unit: participants]
  <65 | 24 | 32 | 21 | 77
  ≥65 | 15 | 24 | 8 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 45 | 26 | 106
  Male | 4 | 11 | 3 | 18
Region of Enrollment [Number; unit: participants]
  United States | 39 | 56 | 29 | 124

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Global Ocular Discomfort Score, Area Under the Curve, Day 0 to Day 28
Description: An electronic Visual Analog Scale (eVAS) was used by the subject to assess ocular discomfort, both frequency and severity, at Day 0 (pre-treatment) and daily thereafter for 28 days. Assessments were entered into a LogPad® (handheld electronic device). The VAS frequency score ranged from 0 (rarely) to 100 (all the time), and the VAS severity score ranged from 0 (very mildly uncomfortable) to 100 (very severely uncomfortable). The Global Ocular Discomfort Score is a composite of the frequency and severity VAS scores (0-100).
Time Frame: Up to 28 days
Population: All subjects randomized to treatment and receiving at least 1 administration of study medication (intent-to-treat). Mixed model repeated measure (MMRM) approach was used to handle missing data during randomized treatment period.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale x days
Groups:
- ESBA105: ESBA105 ophthalmic solution
- Vehicle: ESBA105 vehicle
Arm/Group | ESBA105 | Vehicle
Number analyzed (Participants) | 56 | 29
Units on a scale x days | 63.8773 (2.4832) | 70.2194 (2.39802)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: The safety population includes all subjects exposed to product. Individual subject adverse events, solicited and unsolicited, were collected from time of first instillation of test article (Run-In) until the subject exited the study.
Groups:
- Run-In: ESBA105 vehicle, all participants
Arm/Group | Run-In | ESBA105 | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/56 | 0/29
Other Adverse Events (participants affected / at risk) | 0/124 | 0/56 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.